CLINICAL TRIAL: NCT03887182
Title: Contribution of Functional MRI in Assessment of Auditory Processing Disorders
Acronym: IRMf-TTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP180679; 2018-A03239 (Other: ID-RCB)
Record Dates: First submitted 2019-02-12; First posted 2019-03-22 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2022-07

CONDITIONS: Auditory Processing Disorders
Keywords: auditory processing disorders; functional MRI
MeSH Terms: conditions — Auditory Perceptual Disorders | interventions — Magnetic Resonance Imaging; Exome Sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- confirmed auditory processing disorders (Experimental): functional MRI, Cortical Brainstem Auditory Evoked Potential, Genetic
  Interventions: Diagnostic Test: functional MRI; Diagnostic Test: Automated Cortical Brainstem Auditory Evoked Potential; Genetic: whole exome sequencing
- suspected not confirmed auditory processing disorders (Experimental): functional MRI, Cortical Brainstem Auditory Evoked Potential, Genetic
  Interventions: Diagnostic Test: functional MRI; Diagnostic Test: Automated Cortical Brainstem Auditory Evoked Potential
- healthy volunteers (Active Comparator): functional MRI, Cortical Brainstem Auditory Evoked Potential, Genetic, multidisciplinary consultation
  Interventions: Diagnostic Test: functional MRI; Diagnostic Test: Automated Cortical Brainstem Auditory Evoked Potential; Diagnostic Test: Standard Cortical Brainstem Auditory Evoked Potential; Diagnostic Test: multidisciplinary consultation

INTERVENTIONS:
Diagnostic Test: functional MRI — Additional sequence (DTI) and functional MRI (fMRI) during the MRI which is done as part of the usual care
Diagnostic Test: Automated Cortical Brainstem Auditory Evoked Potential — Automated Cortical Brainstem Auditory Evoked Potential correspond to a non-invasive EEG
Genetic: whole exome sequencing — A study of all the DNA-encoding exons of the child/parent from a sample taken as part of the usual care
  Arms: confirmed auditory processing disorders
Diagnostic Test: Standard Cortical Brainstem Auditory Evoked Potential — Standard Cortical Brainstem Auditory Evoked Potential correspond to a non-invasive EEG
  Arms: healthy volunteers
Diagnostic Test: multidisciplinary consultation — multidisciplinary consultation is composed of:
  * an ENT consultation and audiometry
  * a speech therapy assessment
  * a psychometric evaluation
  Arms: healthy volunteers

SUMMARY:
Auditory Processing Disorder (APD) affects 0.5-7% of the pediatric population. This disorder is responsible for a child's low hearing ability. The diagnosis of APD is difficult because of polymorphic symptoms possibly entangled with other difficulties (learning, communication, attention ...). There is currently no gold standard in the literature for diagnosing APD. Investigators opened multidisciplinary consultation for the children suspected of APD. The purpose of this study is to analyze the results of the multidisciplinary assessment performed on these children (audiometry, cortical auditory brainstem response (ABR), behavioral assessment, psychometric evaluation, genetic analysis) to the results of functional MRI (fMRI) at rest and in activation. The goal is to find radiological MRI-fMRI markers in these patients that improve the diagnosis of APD.

Investigators will compare the f-MRI results between three groups of children in order to find specific radiological markers of APD :

* group 1 : children diagnosed with an Auditory Processing Disorder (APD)
* group 2 : children suspect of APD
* group 3 : children without APD (controls)

DETAILED DESCRIPTION:
The study will include a multidisciplinary consultation with:

* Targeted behavioral assessment auditory processing disorder (APD): speech-in-noise perception, phonemic identification and discrimination, dichotic listening test, temporal processing tests, Random Gap Detection Threshold (RGDT) test.
* Psychometric assessment: assessment of visual / auditory working memory, visual / auditory attention, study of cognitive functions.
* Ear, Nose, Throat (ENT) examination with otoscopy, tonal and vocal audiometry and ABR recording.
* Genetic analysis
* Cortical auditory evoked potential (AEP) recording, compared with the automatized cortical AEP recording on Hear Lab machine.

The purpose of the study is looking for objective biomarkers of APD:

* Compare EEG results with MRI-fMRI results
* Analyze the cortical maturation of children who are fitted with hearings aids: second record of cortical APD performed one year after the fitting.
* Compare the results after one year between group 1 ( with or without hearing aids) and children from group 2.
* MRI-fMRI : to analyze the flow of perfusion, the DTI sequences, and the blood oxygen level-dependent (BOLD) effect (fMRI)

With this multidisciplinary evaluation, the investigators wish to improve the diagnosis of APD in suspected children by associating clinical, radiological, electro-physiological and genetic criteria.

Better understanding and more accurate diagnosis of APD's will improve the care management of these children.

ELIGIBILITY:
Inclusion Criteria Group 1 & 2: :

* 7 to 18 years old
* selected following multidisciplinary consultation whether the diagnosis is confirmed (group G1) or not (group G2).
* Signed consent of both parents
* Affiliated with a health insurance plan

Inclusion Criteria Group 3:

* 7 to 18 years old
* do not present any known hearing pathology
* Signed consent of both parents
* Affiliated with a health insurance plan

Exclusion Criteria:

* Require general anesthesia for MRI
* Contraindication to MRI
* Hearing aids for more than three months prior to inclusion in the study
* Require sedation specifically for research

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
BOLD effect | up to 4 weeks
  BOLD effect is measured during fMRI and compared between the 3 groups of patients

SECONDARY OUTCOMES:
set disyllabic words (Fournier or Boorsma lists) | up to 4 weeks
  Speech evaluation : set disyllabic words using the Fournier or Boorsma lists (the French equivalent of the. Peabody PBK test), depending on age
RapDys | up to 4 weeks
  Speech evaluation
Random Gap Detection Test (RGDT) | up to 4 weeks
  Speech evaluation
Dichotic listening test | up to 4 weeks
  Speech evaluation
temporal pattern recognition test | up to 4 weeks
  Speech evaluation
Test of Everyday Attention for Children (TEA-Ch test) | up to 4 weeks
  Psychometric evaluation for children aged 7-12 years
Wechsler Intelligence Scale for Children (WISC-V) test | up to 4 weeks
  Psychometric evaluation for children aged 13-18 years
Chromosomal analysis (group 1 only) | up to 12 months
  Genetic analysis
Work Environment Scale (WES) sequencing (group 1 only) | up to 12 months
  Genetic analysis
Measures of P1, N1, P2, N2 waves' Latencies | At inclusion day (visit 1) and at 12 months (group 1 and 2 only)
  Cortical Brainstem Auditory Evoked
Measures of P1, N1, P2, N2 waves' amplitudes | At inclusion day (visit 1) and at 12 months (group 1 an 2 only)
  Cortical Brainstem Auditory Evoked
Infusion Rate (MRI-ASL) | up to 4 weeks
  Infusion Rate (MRI-ASL) is measured during MRI
tractography results (DTI sequence) | up to 4 weeks
  tractography results (DTI sequence) is measured during MRI

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Rouillon, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Necker Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chermak GD, Bamiou DE, Vivian Iliadou V, Musiek FE. Practical guidelines to minimise language and cognitive confounds in the diagnosis of CAPD: a brief tutorial. Int J Audiol. 2017 Jul;56(7):499-506. doi: 10.1080/14992027.2017.1284351. Epub 2017 Feb 28. PMID 28635503
- [Background] Moore DR, Ferguson MA, Edmondson-Jones AM, Ratib S, Riley A. Nature of auditory processing disorder in children. Pediatrics. 2010 Aug;126(2):e382-90. doi: 10.1542/peds.2009-2826. Epub 2010 Jul 26. PMID 20660546
- [Background] Barker MD, Kuruvilla-Mathew A, Purdy SC. Cortical Auditory-Evoked Potential and Behavioral Evidence for Differences in Auditory Processing between Good and Poor Readers. J Am Acad Audiol. 2017 Jun;28(6):534-545. doi: 10.3766/jaaa.16054. PMID 28590897
- [Background] Tomlin D, Rance G. Maturation of the Central Auditory Nervous System in Children with Auditory Processing Disorder. Semin Hear. 2016 Feb;37(1):74-83. doi: 10.1055/s-0035-1570328. PMID 27587924
- [Background] Sharma M, Purdy SC, Kelly AS. Comorbidity of auditory processing, language, and reading disorders. J Speech Lang Hear Res. 2009 Jun;52(3):706-22. doi: 10.1044/1092-4388(2008/07-0226). Epub 2008 Dec 8. PMID 19064904
- [Background] de Wit E, Visser-Bochane MI, Steenbergen B, van Dijk P, van der Schans CP, Luinge MR. Characteristics of Auditory Processing Disorders: A Systematic Review. J Speech Lang Hear Res. 2016 Apr 1;59(2):384-413. doi: 10.1044/2015_JSLHR-H-15-0118. PMID 27082630
- [Background] Demanez L, Dony-Closon B, Lhonneux-Ledoux E, Demanez JP. Central auditory processing assessment: a French-speaking battery. Acta Otorhinolaryngol Belg. 2003;57(4):275-90. PMID 14714945
- [Background] Sharma A, Kraus N, McGee TJ, Nicol TG. Developmental changes in P1 and N1 central auditory responses elicited by consonant-vowel syllables. Electroencephalogr Clin Neurophysiol. 1997 Nov;104(6):540-5. doi: 10.1016/s0168-5597(97)00050-6. PMID 9402896
- [Background] Sharma A, Dorman MF, Spahr AJ. Rapid development of cortical auditory evoked potentials after early cochlear implantation. Neuroreport. 2002 Jul 19;13(10):1365-8. doi: 10.1097/00001756-200207190-00030. PMID 12151804
- [Background] Sharma A, Martin K, Roland P, Bauer P, Sweeney MH, Gilley P, Dorman M. P1 latency as a biomarker for central auditory development in children with hearing impairment. J Am Acad Audiol. 2005 Sep;16(8):564-73. doi: 10.3766/jaaa.16.8.5. PMID 16295243
- [Background] Sharma A, Glick H, Campbell J, Biever A. CENTRAL AUDTIORY DEVELOPMENT IN CHILDREN WITH HEARING LOSS: CLINICAL RELEVANCE OF THE P1 CAEP BIOMARKER IN HEARING-IMPAIRED CHILDREN WITH MULTIPLE DISABILITIES. Hearing Balance Commun. 2013 Sep;11(3):10.3109/21695717.2013.812378. doi: 10.3109/21695717.2013.812378. PMID 24273704
- [Background] Sharma M, Purdy S C, Kelly A S. The contribution of speech-evoked cortical auditory evoked potentials to the diagnosis and measurement of intervention outcomes in children with auditory processing disorder. Semin Hear. 2014;35(1):51-64
- [Background] Purdy SC, Kelly AS, Davies MG. Auditory brainstem response, middle latency response, and late cortical evoked potentials in children with learning disabilities. J Am Acad Audiol. 2002 Jul-Aug;13(7):367-82. PMID 12199513
- [Background] Anderson S, Chandrasekaran B, Yi HG, Kraus N. Cortical-evoked potentials reflect speech-in-noise perception in children. Eur J Neurosci. 2010 Oct;32(8):1407-13. doi: 10.1111/j.1460-9568.2010.07409.x. PMID 20950282
- [Background] Cunningham J, Nicol T, Zecker S, Kraus N. Speech-evoked neurophysiologic responses in children with learning problems: development and behavioral correlates of perception. Ear Hear. 2000 Dec;21(6):554-68. doi: 10.1097/00003446-200012000-00003. PMID 11132782
- [Background] Punch S, Van Dun B, King A, Carter L, Pearce W. Clinical Experience of Using Cortical Auditory Evoked Potentials in the Treatment of Infant Hearing Loss in Australia. Semin Hear. 2016 Feb;37(1):36-52. doi: 10.1055/s-0035-1570331. PMID 27587921
- [Background] Martin BA, Tremblay KL, Korczak P. Speech evoked potentials: from the laboratory to the clinic. Ear Hear. 2008 Jun;29(3):285-313. doi: 10.1097/AUD.0b013e3181662c0e. PMID 18453883
- [Background] Micallef LA. Auditory Processing Disorder (APD): Progress in Diagnostics So Far. A Mini-Review on Imaging Techniques. J Int Adv Otol. 2015 Dec;11(3):257-61. doi: 10.5152/iao.2015.1009. PMID 26915160
- [Background] Owen JP, Marco EJ, Desai S, Fourie E, Harris J, Hill SS, Arnett AB, Mukherjee P. Abnormal white matter microstructure in children with sensory processing disorders. Neuroimage Clin. 2013 Jun 23;2:844-53. doi: 10.1016/j.nicl.2013.06.009. eCollection 2013. PMID 24179836
- [Background] Kim MJ, Jeon HA, Lee KM, Son YD, Kim YB, Cho ZH. Neuroimaging features in a case of developmental central auditory processing disorder. J Neurol Sci. 2009 Feb 15;277(1-2):176-80. doi: 10.1016/j.jns.2008.10.020. Epub 2008 Dec 6. PMID 19058816
- [Background] Belin P, Zatorre RJ, Lafaille P, Ahad P, Pike B. Voice-selective areas in human auditory cortex. Nature. 2000 Jan 20;403(6767):309-12. doi: 10.1038/35002078. PMID 10659849
- [Background] Thomsen T, Rimol LM, Ersland L, Hugdahl K. Dichotic listening reveals functional specificity in prefrontal cortex: an fMRI study. Neuroimage. 2004 Jan;21(1):211-8. doi: 10.1016/j.neuroimage.2003.08.039. PMID 14741658
- [Background] Pluta A, Wolak T, Czajka N, Lewandowska M, Ciesla K, Rusiniak M, Grudzien D, Skarzynski H. Reduced resting-state brain activity in the default mode network in children with (central) auditory processing disorders. Behav Brain Funct. 2014 Sep 26;10(1):33. doi: 10.1186/1744-9081-10-33. PMID 25261349
- [Background] Bartel-Friedrich S, Broecker Y, Knoergen M, Koesling S. Development of fMRI tests for children with central auditory processing disorders. In Vivo. 2010 Mar-Apr;24(2):201-9. PMID 20363995